CLINICAL TRIAL: NCT06835075
Title: Clinicaly Manifested Reinfections with Borrelia Burgdorferi Sensu Lato
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Petra Bogovič, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: 0120-551/2023/3
Record Dates: First submitted 2025-01-31; First posted 2025-02-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Lyme Borreliosis
Keywords: Lyme borreliosis; Reinfection; Borrelia burgdorferi sensu lato
MeSH Terms: conditions — Lyme Disease; Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Data on reinfections with B. burgdorferi sensu lato in humans are scarce; they are limited to case reports and a few small groups of patients, mostly from the USA and less frequently from Europe. In these reports, the clinical manifestation of reinfection was usually erythema migrans and was most often documented after successful treatment of a previous infection (almost always erythema migrans). The clinical manifestations of Lyme disease in reinfection appear to be similar to those of primary infection, but there are no studies on possible differences in serological or immunological responses.

The current study has 3 primary objectives:

* To determine the frequency of clinically detectable reinfections and to identify the circumstances under which they occur;
* To determine possible differences between primary and reinfection in clinical presentation, disease course and outcome, and specific serum antibody response;
* To determine the aetiology of clinically detectable reinfections by comparing Borrelia isolates recovered from the skin of the same patient at primary and reinfection.

DETAILED DESCRIPTION:
The current study will encompass all patients aged ≥18 years who were treated at the Department of Infectious Diseases, UMC Ljubljana for proven, clinically well-defined Lyme borreliosis in the period 1989 - 2023. Organised data collection in patients with Lyme borreliosis started in 1986 when we established an Outpatient Lyme borreliosis Clinic and introduced uniform approaches to diagnosis, treatment and follow-up of the disease course, thus obtaining a database of high quality clinical and laboratory data in a large number of patients.

The aims:

1. To determine the frequency of clinically detectable reinfections and to identify the circumstances under which they occur (in a cohort of ~15000 European patients with erythema migrans and ~1500 patients with early extradermal or late Lyme disease).
2. To determine possible differences between primary and reinfection in clinical presentation, disease course and outcome, and specific serum antibody response (by comparing clinical findings and serological test results in ~1500 patients who were diagnosed with erythema migrans more than 1 time).
3. To determine the aetiology of clinically detectable reinfections by comparing Borrelia isolates recovered from the skin of the same patient at primary and reinfection (~100 patients and 200 isolates, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definitive Lyme borreliosis

Exclusion Criteria:

* /

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with definitive Lyme borreliosis at LBOC in the period 35 years (1989 to 2023).
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The frequency of clinically detectable reinfections and identification of the circumstances under which they occur | At diagnosis
Differences between primary erythema migrans and erythema migrans as a result of reinfection according to clinical findings, the presence of borrelial antibodies, and Borrelia skin culture results | The time frame between primary EM and EM as a result of reinfection ranges from 1 month to 35 years.
  The objectives of the current study were to assess and compare findings in patients with primary erythema migrans (EM) skin lesion versus those with EM due to reinfection, including:
  i) clinical findings: age (years), sex, tick bite at the site of EM, duration of EM till diagnosis (days), largest diameter of EM at diagnosis (cm), ring-like EM, number of EM, local symptoms (present or absent), systemic symptoms, underlying chronic illness, abnormalities on physical examination; ii) Borrelia antibody responses (IgM ang IgG determined with chemi-luminescence immunoassay, LIAISON, Diasorin, Saluggia, Italy); iii) Borrelia skin culture positivity rate.
Comparison of the aetiology of clinically detectable reinfections by comparing Borrelia isolates recovered from the skin of the same patient at primary infection and reinfection | The time frame between primary EM and EM as a result of reinfection ranges from 1 month to 35 years.
  1. We will compare the proportion of positive cultures in patients with a primary cutaneous lesion of EM versus patients with EM due to reinfection.
  2. In the subgroup of patients in whom Borrelia were isolated from skin of primary as well as from EM as a result of reinfection, we will compare Borrelia pairs according to species (determined by PCR) and according to sequencing findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
Personal, highly confidential data